CLINICAL TRIAL: NCT04654325
Title: Prevalence of SARS-CoV-2 Genome in Tears of Asymptomatic and Moderately Symptomatic COVID-19 Patients
Acronym: COVIDEYE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: less covid testing
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP201268; 2020-A02996-33 (Other: ID-RCB)
Record Dates: First submitted 2020-11-30; First posted 2020-12-04 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: SARS-CoV-2
Keywords: SARS-CoV-2; COVID19; conjunctiva; tears
MeSH Terms: conditions — COVID-19; Lacerations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients attending to the COVID19 screening facility (Other): Patients will have both nasopharyngeal and conjunctival swab for SARS-CV-2 genome detection using PCR. Study will evaluate the prevalence of positive conjunctival swabs in patients with positive nasopharyngeal swab. These results will be corelated to symptoms of disease assessed with a stan
  Interventions: Diagnostic Test: conjunctival swab

INTERVENTIONS:
Diagnostic Test: conjunctival swab — Patients will have conjunctival swab for SARS-CV-2 genome detection

SUMMARY:
To evaluate the prevalence of SARS-CoV-2 genome in patients with asymptomatic and moderately symptomatic COVID19.

DETAILED DESCRIPTION:
Patients attending to the COVID19 screening facility of Paris South University hospital and willing to participate to the study will have both nasopharyngeal and conjunctival swab for SARS-CV-2 genome detection using PCR. The project will evaluate the prevalence of positive conjunctival swabs in patients with positive nasopharyngeal swab. These results will be corelated to symptoms of disease assessed with a standardized questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving diagnostic nasopharyngeal PCR for COVID-19 as part of the usual care
* Age ≥ 18.
* Information and signature of consent
* Affiliated with a social security scheme or entitled

Exclusion Criteria:

* Refusal to participate in the study
* Eye surgery less than 3 months old
* Unable to give informed consent
* No coverage through the health insurance system
* Patient under judicial protection
* Patient on AME

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
presence of SARS-CoV-2 genome in tears | at the end of the study, an average of 1 year
  Prevalence of SARS-CoV-2 genome in tears

SECONDARY OUTCOMES:
presence of systemic symptoms evaluated at the time of making an appointment by a systematic standardized interrogation | at the end of the study, an average of 1 year
  correlation between systemic symptoms (fever, chills, sweating, muscle aches, headache, runny or stuffy nose, cough, sore throat, asthenia, anosmia, agueusia, unusual shortness of breath, skin rash diarrhea, nausea vomiting) and positive conjunctival swab
assessement of viral load levels | at the end of the study, an average of 1 year
  correlation between nasopharyngeal viral load and conjunctival load (indirectly assessed with cycle thresholds quantification method)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Rousseau, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bicêtre, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No